CLINICAL TRIAL: NCT03144518
Title: A Feasibility Trial of a Brief Positive Affect Intervention to Improve the Effectiveness of Influenza Vaccine Response in Older Adults.
Brief Title: Mood and Influenza Vaccine Response: A Feasibility Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Collaborators: Northumbria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 17039
Record Dates: First submitted 2017-04-28; First posted 2017-05-08 (Actual); Results first posted 2019-07-15 (Actual); Last update posted 2019-07-15 (Actual); Status verified 2019-04

CONDITIONS: Vaccination; Infection
Keywords: Positive Affect; Positive Mood; Influenza Vaccination; Vaccination; Randomised Controlled Trial
MeSH Terms: conditions — Infections; Influenza, Human | interventions — Parturition

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Participants in the experimental condition will view a video designed to induce positive affect. This includes 3 short comedy clips (fork handles sketch, the two Ronnie's; A room with a view - faulty towers; Tim Vine Live stand-up extract), uplifting music (Jailhouse Rock - Elvis Presley; Happy Together - The Turtles), jokes and positive imagery. The content of the intervention has been informed by patient and public involvement, focus groups with older adults, and pilot testing.
  Interventions: Other: Positive Affect Intervention; Biological: Northern Hemisphere Influenza Vaccine 2017/18 (Delivered as part of Standard Care)
- Active Control (Active Comparator): Participants in the control condition will view a video of matched length to the experimental condition video, but not designed to induce mood change. This includes short documentary clips (a pride in pencils; model railways, lecture extract on hydration), neutral music and images.
  Interventions: Other: Neutral Control Intervention; Biological: Northern Hemisphere Influenza Vaccine 2017/18 (Delivered as part of Standard Care)

INTERVENTIONS:
Other: Positive Affect Intervention — See Previous Description
  Arms: Experimental
Other: Neutral Control Intervention — See Previous Description
  Arms: Active Control
Biological: Northern Hemisphere Influenza Vaccine 2017/18 (Delivered as part of Standard Care) — Northern Hemisphere Influenza Vaccine 2017/18 (Delivered as part of Standard Care)

SUMMARY:
This study is a 2-arm, parallel, randomised controlled feasibility trial of a brief video intervention designed to induce positive affect (mood) in older adults in primary care settings prior to the receipt of influenza vaccination. Participants will be randomised into two conditions: experimental and active control. In the experimental condition, participants will view the approximately 15 minute long intervention video immediately prior to vaccination. In the active control condition, participants will view a matched video that is designed to be mood neutral. Pre-and-post positive affect levels will be assessed by self-report questionnaires. Immune response to the intervention and vaccination responses will be assessed in saliva and serum samples respectively.

The objectives of the study are to assess the impact of the intervention on mood, immune function, and antibody response to influenza vaccination in older adults. This feasibility trial will also allow data collection on exploring recruitment, attrition, intervention engagement, and practicality of collecting clinical data available through electronic records to inform the design of a future definitive trial.

DETAILED DESCRIPTION:
The Centers for Disease Control (CDC) describe vaccinations as among the 10 most significant health achievements ever documented; and for many conditions they have been an unmitigated success (e.g., smallpox). There are, however, several populations in whom vaccine effectiveness is far from optimal. These populations are typically contending with underlying immune impairment by virtue of their advancing age and/or the presence of co-existing diseases (e.g., cancer). As a consequence, vaccines are most likely to fail those whom they most seek to benefit: individuals at the greatest risk of ill health.

This has prompted research into treatments that enhance immune function prior to vaccination, so called vaccine adjuvants. The aim of such treatments is to optimise the response the immune system makes to the vaccine antigens and, in so doing, increase the likelihood that the vaccine confers protection.

One area in which there has been interest is in the potential for developing psycho-behavioural vaccine adjuvants. There is considerable evidence that psychological and behavioural factors can modulate immunity; with diet, physical activity, stress, affect, sleep and social support all associated with immune response.

The investigators recently conducted a longitudinal observational cohort study of multiple psychological (positive affect, negative affect, stress) and behavioural (physical activity, sleep, diet) influences on short and long-term antibody responses to influenza vaccination in older adults. This identified positive affect as the most influential psycho-behavioural factor on influenza-specific antibody responses, independently predicting both short and long-term antibody responses in the weakest immunogenic strain above and beyond known demographic and clinical determinants. Intriguingly, the investigators also observed preliminary evidence that positive affect on the day of vaccination was more predictive of antibody responses following vaccination than mood measured over the longer period surrounding vaccination. As influenza-specific antibodies are a well-established correlate of protection from serologically and clinically diagnosed influenza incidence, these data suggest that increasing positive affect immediately prior to vaccination could be used as a non-pharmacological vaccine adjuvant.

Through a series of systematic steps, including focus groups and interviews with older adults and health care professionals, the investigators have recently developed a brief, positive affect intervention - designed to improve short-term mood in older adults and be deliverable within primary care. It is hoped this could act as a psycho-behavioural adjuvant to enhance poor responses to influenza vaccination in older adults. Before performing a definitive trial of the intervention's effectiveness, a feasibility trial is needed for number of reasons:

1. To assess whether our intervention can enhance positive affect (mood)
2. To collect information regarding likely recruitment, effect sizes, and attrition rates for informing the necessary size of a larger definitive trial
3. To examine the practicality and acceptability of delivering the intervention in routine primary care settings
4. To explore the feasibility of obtaining outcome data on healthcare usage for a large scale trial (hospitalisation, GP visits for flu-like symptoms from medical records)

In line with the above, the investigators will be conducting a 2-arm, parallel, randomised controlled feasibility trial of a brief video intervention designed to induce positive affect (mood) in older adults in primary care settings prior to the receipt of influenza vaccination. Participants will be randomised into two conditions: experimental and active control. In the experimental condition, participants will view the approximately 15 minute long intervention video immediately prior to vaccination. In the active control condition, participants will view a matched video that is designed to be mood neutral. Pre-and-post positive affect levels will be assessed by self-report questionnaires. Immune response to the intervention and vaccination responses will be assessed in saliva (pre/post intervention) and serum samples (pre/4 weeks post-vaccination/16weeks post-vaccination) respectively.

ELIGIBILITY:
Inclusion Criteria:

* Males and Females aged 65-85 years (inclusive)
* Received influenza vaccination for the 2016/17 season
* Eligible to receive 2017/18 influenza vaccination as part of usual care
* Ability to give informed consent

Exclusion Criteria:

* Males and Females aged less than 65 or over 85 years (exclusive)
* Did not receive influenza vaccination for the 2016/17 season
* Ineligible to receive 2017/18 influenza vaccination as part of usual care
* Unable to provide informed consent

Deemed by health care provider to be:

* Too physically frail to participate
* Diagnosed with dementia or other cognitive condition which would make participation difficult
* Insufficient command of English language
* Influenza vaccination contraindicated
* Sufficiently impaired of hearing or vision that exposure to the intervention or control video content as intended would be compromised
* Those for whom the collection of blood samples is contraindicated.

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 106 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2017-11-01 (Actual); Study Completion 2018-05-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Nottingham, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Andre FE, Booy R, Bock HL, Clemens J, Datta SK, John TJ, Lee BW, Lolekha S, Peltola H, Ruff TA, Santosham M, Schmitt HJ. Vaccination greatly reduces disease, disability, death and inequity worldwide. Bull World Health Organ. 2008 Feb;86(2):140-6. doi: 10.2471/blt.07.040089. PMID 18297169
- [Background] Jefferson T, Smith S, Demicheli V, Harnden A, Rivetti A, Di Pietrantonj C. Assessment of the efficacy and effectiveness of influenza vaccines in healthy children: systematic review. Lancet. 2005 Feb 26-Mar 4;365(9461):773-80. doi: 10.1016/S0140-6736(05)17984-7. PMID 15733718
- [Background] Calder PC, Jackson AA. Undernutrition, infection and immune function. Nutr Res Rev. 2000 Jun;13(1):3-29. doi: 10.1079/095442200108728981. PMID 19087431
- [Background] Simpson R, Spielmann G. Exercise and Immunosenescence. In: Bosch J, Phillips A, Lord J, eds. Immunosenescence. New York: : Springer Science 2013. 159-78.
- [Background] Centers for Disease Control and Prevention (CDC). Ten great public health achievements--worldwide, 2001-2010. MMWR Morb Mortal Wkly Rep. 2011 Jun 24;60(24):814-8. PMID 21697806
- [Background] Segerstrom SC, Miller GE. Psychological stress and the human immune system: a meta-analytic study of 30 years of inquiry. Psychol Bull. 2004 Jul;130(4):601-30. doi: 10.1037/0033-2909.130.4.601. PMID 15250815
- [Background] Pressman SD, Cohen S. Does positive affect influence health? Psychol Bull. 2005 Nov;131(6):925-971. doi: 10.1037/0033-2909.131.6.925. PMID 16351329
- [Background] Bryant PA, Trinder J, Curtis N. Sick and tired: Does sleep have a vital role in the immune system? Nat Rev Immunol. 2004 Jun;4(6):457-67. doi: 10.1038/nri1369. No abstract available. PMID 15173834
- [Background] Uchino BN. Social support and health: a review of physiological processes potentially underlying links to disease outcomes. J Behav Med. 2006 Aug;29(4):377-87. doi: 10.1007/s10865-006-9056-5. Epub 2006 Jun 7. PMID 16758315
- [Background] Coudeville L, Bailleux F, Riche B, Megas F, Andre P, Ecochard R. Relationship between haemagglutination-inhibiting antibody titres and clinical protection against influenza: development and application of a bayesian random-effects model. BMC Med Res Methodol. 2010 Mar 8;10:18. doi: 10.1186/1471-2288-10-18. PMID 20210985
- [Derived] Ayling K, Fairclough L, Buchanan H, Wetherell MA, Vedhara K. Mood and influenza vaccination in older adults: A randomized controlled trial. Health Psychol. 2019 Nov;38(11):984-996. doi: 10.1037/hea0000786. Epub 2019 Aug 5. PMID 31380684

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Note: 3 Participants were not randomised to condition, as they did not attend primary session.
Period: Primary Outcome (Mood)
Arm/Group | Experimental | Active Control
Started | 52 | 51
Completed | 52 | 51
Not Completed | 0 | 0
Period: 4 Weeks Post-Vaccination
Arm/Group | Experimental | Active Control
Started | 52 | 51
Completed | 51 | 51
Not Completed | 1 | 0
Period: 16 Week Post-Vaccination
Arm/Group | Experimental | Active Control
Started | 52 | 51
Completed | 49 | 49
Not Completed | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental | Active Control | Total
Number analyzed (Participants) | 52 | 51 | 103
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Missing Data count n=1
  years
    number analyzed (Participants) | 52 | 50 | 102
    (all) | 72.6 (4.6) | 73.3 (5.1) | 72.95 (4.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 30 | 52
  Male | 30 | 21 | 51
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 51 | 48 | 99
  Asian | 0 | 1 | 1
  Black | 1 | 1 | 2
  Did not Respond | 0 | 1 | 1
Marital Status [Count of Participants; unit: Participants]
  Married | 34 | 29 | 63
  Single, never married | 0 | 3 | 3
  Separated/divorced | 9 | 4 | 13
  Widowed | 4 | 8 | 12
  Cohabiting | 3 | 3 | 6
  Did not Respond | 2 | 4 | 6
Highest Level of Education [Count of Participants; unit: Participants]
  School | 37 | 40 | 77
  Undergraduate | 2 | 0 | 2
  Postgraduate | 0 | 1 | 1
  Other | 8 | 8 | 16
  Did not respond | 5 | 2 | 7
Independent Living [Count of Participants; unit: Participants]
  Yes | 47 | 49 | 96
  No | 5 | 2 | 7
Highest Ever Total Household Income [Count of Participants; unit: Participants]
  ≤ £14,999 | 17 | 16 | 33
  £15,000-£24,999 | 16 | 17 | 33
  £25,000-£34,999 | 8 | 4 | 12
  £35,000-£49,000 | 7 | 5 | 12
  £50,000-£74,999 | 1 | 2 | 3
  £75,000-£99,000 | 0 | 0 | 0
  ≥ £100,000 | 0 | 0 | 0
  Did Not Respond | 3 | 7 | 10
Current Smoker [Count of Participants; unit: Participants] | 4 | 4 | 8
Total Health Status [Mean (Standard Deviation); unit: units on a scale] — Health Status Questionnaire 2.0 (Barry, Kaiser, & Atwood, 2007). Responses are weighted and summed as per published guidelines in above reference to calculate a total perceived health status score ranging from a minimum of 0 to a maximum of 800, with higher scores indicating greater perceived health. Population: Missing Data Count: n=6
  units on a scale
    number analyzed (Participants) | 49 | 48 | 97
    (all) | 555.7 (175.1) | 555.1 (169.9) | 555.41 (171.62)
Trait Positive Affect [Mean (Standard Deviation); unit: units on a scale] — Trait positive affect was measured using positive affect sub scale from the Positive and Negative Affect Schedule (Watson et al., 1988). Positive subscale (α = .92) was created by summing the scores of positive adjectives. Minimum score 10, Maximum Score 50, with higher scores indicating greater trait positive affect. Population: Missing Data Count: n=8
  units on a scale
    number analyzed (Participants) | 50 | 45 | 95
    (all) | 33.5 (8.6) | 33.8 (8.1) | 33.65 (8.33)
Trait Optimism [Mean (Standard Deviation); unit: units on a scale] — Trait optimism was measured using the Revised Life Orientation Test (Scheier, Carver, & Bridges, 1994). Six items are used to compute a trait optimism score (α = .73) in line with published guidelines. Minimum Score 0, Maximum Score 24 with higher scores indicating with greater optimism. Population: Missing Data Count: n=7
  units on a scale
    number analyzed (Participants) | 50 | 46 | 96
    (all) | 16.0 (4.8) | 15.3 (4.5) | 15.68 (4.61)
Trait Emotional Reactivity [Mean (Standard Deviation); unit: units on a scale] — Trait emotional reactivity was measured using the 21-item Emotional Reactivity Scale (Nock, Wedig, Holmberg, & Hooley, 2008). Items scores are summed (α = .96). Minimum score 21, maximum score 105, with greater scores indicating greater trait emotional reactivity. Population: Missing Data Count: n=8
  units on a scale
    number analyzed (Participants) | 47 | 48 | 95
    (all) | 39.9 (17.2) | 41.3 (16.0) | 40.59 (16.52)
Pre-Vaccination IgG [Mean (Standard Deviation); unit: ug/ml] — Values represent equivalent ug/ml based on diluted sample absorbance value interpolation against a standard IgG curve, multiplied by the serum dilution score (i.e., 4000).
  ug/ml
    A/Michigan | 187.2 (112.4) | 156.6 (103.1) | 172.05 (108.47)
    A/Hong-Kong | 238.0 (119.9) | 241.0 (158.1) | 239.50 (139.42)
    B/Brisbane | 107.0 (54.1) | 118.9 (78.7) | 112.90 (67.35)
    B/Phuket | 144.4 (85.1) | 183.2 (146.2) | 163.61 (117.93)
Trait Negative Affect [Mean (Standard Deviation); unit: units on a scale] — Trait negative affect was measured using the negative affect sub scale of Positive and Negative Affect Schedule (Watson et al., 1988). Negative affect subscales (α = .92) was created by summing the scores of negative adjectives. Minimum score 10, maximum score 50 with higher scores indicating greater trait negative affect. Population: Missing Data Count n=11
  units on a scale
    number analyzed (Participants) | 49 | 43 | 92
    (all) | 15.2 (6.7) | 15.5 (6.4) | 15.35 (6.52)

OUTCOME MEASURES:

1. Primary Outcome: Mood Outcome Scores [Multiple]
Description: Affective Slider (Betella & Verschure, 2016), consists of two single item visual analogue scales. Scores for each are presented as a value from 0 to 100 with higher scores indicating greater pleasure (VAS-Valence) and arousal (VAS-Arousal).
  Positive and Negative Affect Schedule (Watson et al., 1988). Positive and negative affect subscales were created by summing the scores of positive and negative adjectives respectively. For each sub scale, minimum score = 10, maximum score = 50 with higher scores indicating greater positive and negative affect respectively.
  Pictorial scale of positive affect (unvalidated, internally developed). Participants completed a single-item photo-based measure of positive affect tailored for older adults. Participants were presented with six groups of images depicting varying degrees of positive affect, and indicate which best reflected how they felt at that moment. Minumum score 1, maximum score 6, higher scores indicate greater positive affect.
Time Frame: Baseline, Immediately Post Intervention (i.e, 15 minutes post-baseline).
Population: Missing Data for some outcome measures - i.e., incomplete scale
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental | Active Control
Number analyzed (Participants) | 52 | 51
score on a scale
  Post-Intervention VAS-Valence | 87.4 (15.7) | 79.8 (20.8)
  Post-Intervention VAS-Arousal | 83.7 (16.8) | 79.8 (20.3)
  Post-Intervention Pictorial Scale: number analyzed (Participants) | 50 | 51
  Post-Intervention Pictorial Scale | 4.7 (1.1) | 4.0 (1.5)
  Post-Intervention PANAS Positive Affect: number analyzed (Participants) | 52 | 49
  Post-Intervention PANAS Positive Affect | 35.0 (8.4) | 35.0 (7.6)
  Post-Intervention PANAS Negative Affect | 11.1 (3.0) | 11.4 (2.3)
  Pre-Intervention VAS-Valence: number analyzed (Participants) | 49 | 51
  Pre-Intervention VAS-Valence | 79.5 (19.2) | 80.5 (18.1)
  Pre-Intervention VAS-Arousal: number analyzed (Participants) | 49 | 51
  Pre-Intervention VAS-Arousal | 79.9 (19.0) | 80.9 (20.1)
  Pre-Intervention Pictorial: number analyzed (Participants) | 50 | 49
  Pre-Intervention Pictorial | 3.7 (1.5) | 4.0 (1.5)
  Pre-Intervention PANAS Postive Affect | 34.3 (7.2) | 34.6 (35.0)
  Pre-Intervention PANAS Negative Affect | 12.3 (4.0) | 12.3 (4.0)
Statistical Analysis 1: Comparison: Experimental vs Active Control; VAS-Valence Scores; Test type: Superiority; p = .005, ANCOVA — ANCOVA, controlling for pre-intervention levels; ANCOVA, controlling for pre-intervention levels; Partial Eta Squared = .079, 90% CI 2-sided [.014 to .173]
Statistical Analysis 2: Comparison: Experimental vs Active Control; VAS-Arousal Scores; Test type: Superiority; p = .047, ANCOVA; Controlling for pre-intervention scores; Partial Eta-Squared = .04, 90% CI 2-sided [.000 to .120]
Statistical Analysis 3: Comparison: Experimental vs Active Control; Pictorial Scale; Test type: Superiority; p = .002, ANCOVA; Controlling for pre-intervention levels; Partial Eta Squared = .096, 90% CI 2-sided [.022 to .196]
Statistical Analysis 4: Comparison: Experimental vs Active Control; PANAS Positive Affect Scores; Test type: Superiority; p = .697, ANCOVA; Controlling for baseline levels; Partial Eta Squared = .002, 90% CI 2-sided [.000 to .036]
Statistical Analysis 5: Comparison: Experimental vs Active Control; PANAS Negative Affect Scores; Test type: Superiority; p = .462, ANCOVA; Partial Eta Squared = .005, 90% CI 2-sided [.000 to .053]

2. Secondary Outcome: Recruitment
Description: Recruitment rates to inform a future definitive trial
Time Frame: Baseline
Population: Total Population that received study Invitation
Measure: Count of Participants; unit: Participants
Groups:
- Whole Trial: Recruitment Details are presented for trial as a whole
Arm/Group | Whole Trial
Number analyzed (Participants) | 1131
Participants
  Expressed Interest, but not consented | 23
  Consented, but not randomised | 3
  Randomised | 103
  Did Not Express Interest | 1002

3. Secondary Outcome: Attrition
Description: Attrition - to inform a future definitive trial
Time Frame: 4 weeks (post-vaccination), 16 Weeks (post-vaccination)
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental | Active Control
Number analyzed (Participants) | 52 | 51
Participants
  Attendance at 4 Week Follow-up: Yes | 51 | 51
  Attendance at 4 Week Follow-up: No | 1 | 0
  Attendance at 16 Week Follow up: Yes | 49 | 48
  Attendance at 16 Week Follow up: No | 3 | 3

4. Secondary Outcome: Secretory IgA Response
Description: Secretory IgA levels measured in saliva samples via ELISA. This is a non-specific measure of immunological response
Time Frame: Baseline, Immediately Post Intervention (i.e, 15 minutes post-baseline).
Population: Missing Data Count n=15
Measure: Mean (Standard Deviation); unit: Flow Rate (ug/min)
Arm/Group | Experimental | Active Control
Number analyzed (Participants) | 46 | 42
Flow Rate (ug/min)
  Pre-Intervention Flow Rate | 81.0 (76.4) | 94.1 (94.2)
  Post-Intervention Flow Rate: number analyzed (Participants) | 46 | 41
  Post-Intervention Flow Rate | 116.7 (107.5) | 144.7 (142.5)
Statistical Analysis 1: Comparison: Experimental vs Active Control; Test type: Superiority; p = .806, ANCOVA; Controlling for pre-intervention levels; Partial Eta Squared = .001, 90% CI 2-sided [.000 to .031]

5. Secondary Outcome: Vaccine Specific IgG Response
Description: IgG levels against the 4 vaccine strains measured via ELISA.
  Values represent equivalent ug/ml based on diluted sample absorbance value interpolation against a standard IgG curve, multiplied by the serum dilution score (i.e., 4000).
Time Frame: 4 weeks (post-vaccination), 16 Weeks (post-vaccination)
Population: Missing Data Count: n=1 for 4 weeks post-vaccination, n=5 for 16 weeks post-vaccination
Measure: Mean (Standard Deviation); unit: ug/ml
Arm/Group | Experimental | Active Control
Number analyzed (Participants) | 52 | 51
ug/ml
  4 Weeks Post-Vaccination A/Michigan: number analyzed (Participants) | 51 | 51
  4 Weeks Post-Vaccination A/Michigan | 243.28 (134.52) | 208.81 (122.42)
  4 Weeks Post-Vaccination A/Hong-Kind: number analyzed (Participants) | 51 | 51
  4 Weeks Post-Vaccination A/Hong-Kind | 301.68 (138.88) | 284.96 (138.64)
  4 Weeks Post-Vaccination B/Brisbane: number analyzed (Participants) | 51 | 51
  4 Weeks Post-Vaccination B/Brisbane | 126.30 (56.36) | 127.25 (63.93)
  4 Weeks Post-Vaccination B/Phuket: number analyzed (Participants) | 51 | 51
  4 Weeks Post-Vaccination B/Phuket | 210.30 (123.96) | 229.57 (135.63)
  16 Weeks Post-Vaccination A/Michigan: number analyzed (Participants) | 49 | 49
  16 Weeks Post-Vaccination A/Michigan | 221.69 (131.90) | 203.03 (119.41)
  16 Weeks Post-Vaccination A/Hong-Kong: number analyzed (Participants) | 49 | 49
  16 Weeks Post-Vaccination A/Hong-Kong | 283.67 (126.72) | 288.75 (180.18)
  16 Weeks Post-Vaccination B/Brisbane: number analyzed (Participants) | 49 | 49
  16 Weeks Post-Vaccination B/Brisbane | 139.49 (56.40) | 144.47 (76.77)
  16 Weeks Post-Vaccination B/Phuket: number analyzed (Participants) | 49 | 49
  16 Weeks Post-Vaccination B/Phuket | 249.10 (124.90) | 271.70 (176.16)
Statistical Analysis 1: Comparison: Experimental vs Active Control; 4 Weeks A/Hong-Kong; Test type: Superiority — Note: The study was not powered a priori to detect significant differences in these outcomes; p = .438, ANCOVA; Controlling for Pre-Vaccination levels; Partial Eta Squared = .006, 90% CI 2-sided [.000 to .055]
Statistical Analysis 2: Comparison: Experimental vs Active Control; A/Hong-Kong 16 Weeks Post-Vaccination; Test type: Superiority — Note: The study was not powered a priori to detect significant differences in these outcomes; p = .516, ANCOVA; controlling for pre-vaccination levels; Partial Eta Squared = .004, 90% CI 2-sided [.000 to .051]
Statistical Analysis 3: Comparison: Experimental vs Active Control; A/Michigan 4 weeks post-vaccination; Test type: Superiority — Note: The study was not powered a priori to detect significant differences in these outcomes; p = .671, ANCOVA; controlling for pre-vaccination levels; Partial Eta Squared = .002, 90% CI 2-sided [.000 to .038]
Statistical Analysis 4: Comparison: Experimental vs Active Control; A/Michigan 16 weeks post-vaccination; Test type: Superiority — Note: The study was not powered a priori to detect significant differences in these outcomes; p = .980, ANCOVA; Controlling for pre-vaccination levels; Partial Eta Squared = .000, 90% CI 2-sided [.000 to .000]
Statistical Analysis 5: Comparison: Experimental vs Active Control; B/Brisbane 4 weeks post-vaccination; Test type: Superiority — Note: The study was not powered a priori to detect significant differences in these outcomes; p = .409, ANCOVA; Controlling for pre-vaccination levels; Partial Eta Squared = .007, 90% CI 2-sided [.000 to .057]
Statistical Analysis 6: Comparison: Experimental vs Active Control; B/Brisbane 16 weeks post-vaccination; Test type: Superiority — Note: The study was not powered a priori to detect significant differences in these outcomes; p = .377, ANCOVA; Controlling for pre-vaccination levels; Partial Eta Squared = .008, 90% CI 2-sided [.000 to .062]
Statistical Analysis 7: Comparison: Experimental vs Active Control; B/Phuket 4 weeks post-vaccination; Test type: Superiority; p = .892, ANCOVA; Controlling for pre-vaccination levels; Partial Eta Squared = .000, 90% CI 2-sided [.000 to .008]
Statistical Analysis 8: Comparison: Experimental vs Active Control; Test type: Superiority — Note: The study was not powered a priori to detect significant differences in these outcomes; p = .426, ANCOVA; Controlling for pre-vaccination levels; Partial Eta Squared = .007, 90% CI 2-sided [.000 to .058]

6. Secondary Outcome: Health Care Utilization
Description: Via medical records, we assessed health care usage potentially attributable to flu-like symptoms (e.g., GP visits, hospitalisation, antibiotic prescription) during the 6 months post-vaccination
Time Frame: Baseline to 6 months post-vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental | Active Control
Number analyzed (Participants) | 52 | 51
Participants
  GP Consultations | 14 | 13
  Nurse Consultations | 1 | 1
  Out of Hours/Telephone Conversations | 7 | 3
  Emergency Department Consultations | 1 | 1
  Antibiotic Prescriptions | 6 | 9
  Additional Investigations (e.g., Xray) | 4 | 3

ADVERSE EVENTS:
Time Frame: During Primary Study Period - Baseline to 16 weeks post-vaccination.
Arm/Group | Experimental | Active Control
All-Cause Mortality (participants affected / at risk) | 0/52 | 0/51
Serious Adverse Events (participants affected / at risk) | 0/52 | 0/51
Other Adverse Events (participants affected / at risk) | 0/52 | 0/51

LIMITATIONS AND CAVEATS:
The study did not include a usual care comparator. Blinding potentially compromised by common reactions of participants to the positive mood intervention (e.g., laughter). Demand characteristics. Lack of ethnic diversity within sample

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-21): https://cdn.clinicaltrials.gov/large-docs/18/NCT03144518/Prot_SAP_000.pdf